CLINICAL TRIAL: NCT02090556
Title: Long-term Experience With Abatacept SC in Routine Clinical Practice
Acronym: ASCORE
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: inVentiv Health Clinical (Other); PharmaNet (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-348
Record Dates: First submitted 2014-02-19; First posted 2014-03-18 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1:: RA patients naive of Abatacept and any other biologic agents
- Cohort 2:: RA patients naive of Abatacept and who previously failed one or more biologic agents

SUMMARY:
The purpose of this study is to estimate the retention rate of Abatacept SC over 24 months in routine clinical practice, in rheumatoid arthritis patients, in each country involved in the study. The purpose of the UK substudy is to explore whether integrating self-assessment into routine care could maintain tight control (of inflammation/disease activity) and at potentially lower cost resulting in improved health outcomes and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old at treatment initiation
* Patients diagnosed with established moderate to severe active RA as per the 1987 ACR criteria/2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Rheumatoid Arthritis Classification Criteria
* Patients naïve of Abatacept IV and who at their physician's discretion are initiated with Abatacept SC. In countries where required (e.g. Germany and Spain), patients naïve of Abatacept IV and who at their physician's discretion have been initiated with Abatacept SC at least 1 month prior to enrollment visit up to 6 months if baseline and disease characteristics data are available
* For Spanish pharmacogenomic sub-study:
* Caucasian patient and from European ancestry
* Patient for whom a collection of blood sample before the initiation of abatacept is possible or available (blood sample was taken in routine practice before the study enrolment)
* Patient who agreed to participate in this substudy and provide a specific signed Pharmacogenomic Blood RNA informed consent
* In the UK, the ART substudy will be proposed to all patients enrolled in ASCORE from amendment approval and application date

Exclusion Criteria:

- Patients who are currently included in any interventional clinical trial in RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Corhort 1: RA patients naive of Abatacept and any other biologic agents.
  Corhort 2: RA patients naïve of Abatacept and who previously failed one or more biologic agents.
  In Germany, the study will be proposed to patients using syringe or pre-filled pen devices
Sampling Method: Non-Probability Sample
Enrollment: 2954 (Actual)
Dates: Start 2013-03-26 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Key Primary: Median time and estimation of treatment retention rate of Rheumatoid arthritis (RA) patients treated with Abatacept subcutaneous (SC) over 24 months in routine clinical practices | Up to 24 Months
Co-Primary: Description of how Abatacept SC is prescribed in participating countries for each cohort | Up to 24 Months
  Description include concomitant treatments, dosage and adherence to treatment
Co-Primary: Description of the major characteristics of Abatacept SC treated patients (joint population) at treatment initiation | Up to 24 Months
  Major characteristics of population of patients (joint population depending on previous prescriptions) include socio-demographic data, medical history, disease history, co-morbidities and clinical measures
Co-Primary: Impact of the Abatacept SC treatment on health status of each population of patients over time as assessed by morbi-mortality criteria and safety | Up to 24 Months
  Morbi-mortality criteria include clinical measures, Patient Reported Outcomes (PRO) including self-completion quality of life (QoL) questionnaires and healthcare resource use, incidence of local site injection reaction, incidence of long-term adverse events (AE), withdrawal from study due to AE and Serious Adverse Events (SAE)
Co-Primary: Acceptability of the pre-filled pen device based on questionnaires | Up to 24 Months
  Patients using the pre-filled pen will complete questionnaires on overall acceptability of the pre-filled pen device, injection site pain assessment and experience with previous injections

SECONDARY OUTCOMES:
Major determinants of Abatacept SC retention rate | Up to 24 months
  Major determinants including socio-demographic characteristics at treatment initiation, previous biologic treatments, clinical measurements (i.e. Simplified Disease Activity Score based on 28 joints (DAS28), Clinical Disease Activity Index (CDAI), Simple Disease Activity Index (SDAI) and their derived criteria) and PROs such as Health Assessment Questionnaire Disability Index (HAQ-DI) and according to local clinical practices and/or according to local requirements Work Productivity and Activity Impairment Questionnaire:Rheumatoid Arthritis (WPAI:RA), Rheumatoid Arthritis Disease Activity Index (RADAI) or PRO-CLinical Arthritis Activity (PROCLARA) at treatment initiation and/or at studied drug discontinuation
Distribution of time-to-discontinuation of Abatacept SC therapy for each major determinant identified | Up to 24 months
Time to discontinuation of Abatacept (whatever the formulation, SC or IV) | Up to 24 months

OTHER OUTCOMES:
Treatment experience and outcomes after Abatacept discontinuation and switch to a biologic agent or conventional disease modifying anti-rheumatismal drug (DMARD) | Up to 24 months
Build and validate a multigenic predictive model of abatacept clinical response in two different populations of abatacept patients (MTX-IR and anti TNF-IR) (in Spain) | Up to 24 months
Examine how patients self-reporting related to main ASCORE study treatment decisions and explore patients'acceptability of self-monitoring using qualitative methods (ART substudy, in the UK) | Up to 24 months
Patient-reported elements which are most likely to lead to change in therapy (in the UK) | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- Local Institution, Geelong, Victoria, Australia
- Local Institution, Vienna, Austria
- Local Institution, Lille, France
- Local Institution, Dresden, Germany
- Local Institution, Crete, Greece
- Local Institution, Pavia, Italy
- Local Institution, Monaco, Monaco
- Local Institution, Amsterdam, Netherlands
- Local Institution, Barcelona, Spain
- Local Institution, Diessenhofen, Switzerland
- United Kingdom (2):
  - Local Institution, Hull, Yorkshire
  - Local Institution, Cambridgeshire

REFERENCES:
- [Derived] Alten R, Behar C, Merckaert P, Afari E, Vannier-Moreau V, Ohayon A, Connolly SE, Najm A, Juge PA, Liu G, Rai A, Elbez Y, Lozenski K. Predicting abatacept retention using machine learning. Arthritis Res Ther. 2025 Feb 1;27(1):20. doi: 10.1186/s13075-025-03484-0. PMID 39893489
- [Derived] Alten R, Tony HP, Bannert B, Nusslein H, Rauch C, Connolly SE, Chartier M, Lozenski K, Hackl R, Forster A, Peichl P. Subcutaneous abatacept for the treatment of rheumatoid arthritis in routine clinical practice in Germany, Austria, and Switzerland: 2-year retention and efficacy by treatment line and serostatus. Clin Rheumatol. 2023 Sep;42(9):2321-2334. doi: 10.1007/s10067-023-06649-x. Epub 2023 Jun 14. PMID 37314665
- [Derived] Alten R, Mariette X, Flipo RM, Caporali R, Buch MH, Patel Y, Marsal S, Sanmarti R, Nurmohamed MT, Griffiths H, Peichl P, Bannert B, Chartier M, Connolly SE, Lozenski K, Rauch C. Retention of subcutaneous abatacept for the treatment of rheumatoid arthritis: real-world results from the ASCORE study: an international 2-year observational study. Clin Rheumatol. 2022 Aug;41(8):2361-2373. doi: 10.1007/s10067-022-06176-1. Epub 2022 May 10. PMID 35536413
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx